CLINICAL TRIAL: NCT00480233
Title: Validation of a Hebrew Version of a Brief Screening Questionnaire for Depression in General Medicine
Brief Title: Screening Questionnaire for Depression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Raz Gross, Head, Mental Health Epidemiology, The Gertner Institute for Epidemiology
Other Study IDs: SHEBA-06-4420-RG-CTRL
Record Dates: First submitted 2007-05-29; First posted 2007-05-30 (Estimated); Last update posted 2008-02-06 (Estimated); Status verified 2008-02

CONDITIONS: Depression
Keywords: depression; screening; primary care; validity; Hebrew; Primary care and general medical patients
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Depression is common in primary care and general medical settings, but is often unrecognized and untreated by physicians working in those settings.

The Patient Health Questionnaire for depression (PHQ-9) is well validated and widely used screening instrument.

ELIGIBILITY:
Inclusion Criteria:

* >18 yrs
* Primary care and general medical patients
* Understand the IC
* Speaks Hebrew
* No significant cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care and general medical patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-01

CONTACTS AND LOCATIONS:
Overall Officials: Raz Gross, MD, MPH, Principal Investigator — The Gertner Institute
Locations (1):
- Sheba Medical Center and Maccabi Health Services, Tel Litwinsky, Israel